CLINICAL TRIAL: NCT05129956
Title: Efficacy Evaluation of Laparoscopic Sonoguided-microwave Uterine Myoma Ablation
Brief Title: Sonoguided-microwave Uterine Myoma
Acronym: myoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20210131
Record Dates: First submitted 2021-10-28; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: Obstetric/Gynecology
Keywords: microwave; uterine myoma
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- therapy group (Experimental)
  Interventions: Device: "Covidien" Emprint Ablation System with Thermosphere Technology

INTERVENTIONS:
Device: "Covidien" Emprint Ablation System with Thermosphere Technology — The ablation time and wattage are determined according to the size of the tumor. The wattages are respectively 45W, 75W, and 100W, and the maximum time is 10 minutes
  Other Names: "Covidien" Emprint Percutaneous Antenna with Thermosphere Technology

SUMMARY:
This study mainly evaluates the resolution of uterine fibroids by microwave ablation. The medical equipment used is Ke Hui. "The Ampening ablation system is a percutaneous surgery. During laparoscopic surgery, it is directly ablated and soft, including problems that cannot be solved by partial or complete tissue ablation. "Hydrogen is used. If the expected range of ablation can be found, there is no need to wait for 3 to 6 months for ablation slowly like Haifu surgery. A fast, small, high-quality treatment that provides reference for medical treatment and helps doctors choose the most suitable treatment.

DETAILED DESCRIPTION:
A collection of 20 women suffering from uterine fibroids were treated with microwave fibroids ablation for symptoms of uterine fibroids, and they could be discharged the next day or two days after surgery. Schedule return visits and routine blood tests according to clinical needs, and follow up with ultrasound and questionnaires during routine return visits (1, 3, and 6 months) after surgery. In the third month after surgery, there will be another imaging report. Magnetic resonance imaging and blood tests are used to compare the changes of patients' fibroids, their physiological recovery status, and the degree of improvement in their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Women who have reached the age of 20 and have not yet menopause.
2. Myoma size≧4cm.
3. Patients with submucosal fmyoma or intramural myoma of the uterus.

Exclusion Criteria:

1. Patients with subserosal myoma.
2. Pregnant, breastfeeding or have menopause.
3. Pelvic infections, vaginitis, cervicitis or endometritis and have not been cured.
4. Malignant diseases of the cervix and uterus.
5. Abnormal reports of clinical significance in Pap smear or thin-layer cell test.
6. Abnormal blood coagulation function or liver and kidney function, with bleeding tendency.
7. There is no safe puncture treatment route.
8. Those who have installed intrauterine contraceptive device or Pacemaker.
9. Those who cannot perform vaginal ultrasound, such as those who have no sexual experience and do not accept hymen repair.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Uterine myoma ablation | 1 momth
  The ablation range of fibroids can be reduced by 50%, measured by MRI cubic centimeter volume.
Improve bleeding | 3 momths
  The hemoglobin changes before and 3 months after the operation are used to evaluate the improvement of patients' bleeding problems.

SECONDARY OUTCOMES:
Reduce days in hospital | 6 momths
  Reduce the number of hospitalization days for patients to be less than or equal to 4 days.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Yu Long, Professor, Principal Investigator — Department of Obstetrics and Gynecology, Kaohsiung Municipal Hsiao-Kang Hospital, Kaohsiung Medical University, Kaohsiung, Taiwan
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH), Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
The research results are clarified and then set and shared.